CLINICAL TRIAL: NCT06471153
Title: BASNEF Behavioral Transformation: Effect of Empowerment Program on Children's Knowledge, Attitude, Self-Efficacy, and Practice of Nail Biting.
Brief Title: Effect of Empowerment Program on Children's Knowledge, Attitude, Self-Efficacy, and Practice of Nail Biting.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Zohour Ibrahim Mahmoud Rashwan, Assisstant Profesor, Alexandria University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 7/2022PEDI2-1
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Nail Biting
Keywords: BASNEF Model; Children; Knowledge; Nail Biting; Practice; Self-efficacy
MeSH Terms: conditions — Nail Biting

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Received the empowerment program based on the BASNEF model
  Interventions: Behavioral: Empowerment Program Based on BASNEF Model
- Control Group (Active Comparator): received the routine care
  Interventions: Behavioral: Routine Health Education

INTERVENTIONS:
Behavioral: Empowerment Program Based on BASNEF Model — Initially, the researcher established rapport with children of both groups and their gradians, screened them for the eligibility criteria, explained the aim of the study, the duration and nature of the training sessions, and obtained informed assent. The researcher established the session objectives and learning activities and prepared the learning materials. The researchers also prepared the learning environment. The Empowerment program is implemented in accordance with the BANCEF model for behavior transformation into four educational sessions. After the intervention, children's nail-biting knowledge, practice, attitude, and self-efficacy were reassessed.
  Arms: Study Group
Behavioral: Routine Health Education — Children in the control group received routine health education about the problems of nail-biting and routine advice to quit nail-biting.
  Arms: Control Group

SUMMARY:
The study aims to evaluate the effect of an empowerment program based on the BASNEF model on children's knowledge, attitude, self-efficacy, and practice of nail biting.

Research Hypothesis H1: The application of an empowerment program based on the BASNEF model has a positive impact on children's knowledge, attitude, self-efficacy, and practice of nail biting.

DETAILED DESCRIPTION:
Nail-biting or onychophagia is a common phenomenon affecting children where excessive nail-biting is associated with several adverse consequences beyond mere appearance. The aim is to evaluate the effect of an empowerment program based on the BASNEF model on children's knowledge, attitude, self-efficacy, and practice of nail biting.

A quasi-experimental study was conducted in the pediatric wards of Menoufia University Hospital and Benha University Hospital. A convenience sample of 135 children aged 6 to 18 was randomly assigned to two groups. The study group attended four empowerment sessions based on the BANSEF model, emphasizing age-appropriate information, fostering a positive attitude towards quitting nail-biting, discovering the subjective norms that influence nail-biting behaviors, and equipping children with enabling factors to quit. The control group received routine health education.

ELIGIBILITY:
Inclusion Criteria:

* Had nail-biting habits
* Willing to attend the educational sessions

Exclusion Criteria:

* Had history of mental illness

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 135 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Children's Nail-Biting Knowledge | one month
  It includes ten questions about nail biting revolving around the definition (2 items), predisposing factors (2 items), complications and adverse effects (3 items), and management (3 items). A score of (1) was given for the correct answer and zero for the incorrect one.
Children's Nail-Biting Practice/Habits | one month
  It includes ten items describing the children's nail-biting habit, including frequency and duration (2 items), aggravating factors (2 items), areas involved in nail-biting (3 items), and description of nail-biting behavior (3 items). They are instructed to self-monitor their nail-biting behaviors on five a 5-point Likert scale ranging from very frequent (4) to never (0).
Children's Attitude and Self-efficacy Towards Nail-biting | one month
  It consists of 13 items; 10 items measure the child's attitude, and three items assess their intention to act (self-efficacy). Children were asked to rate their answers on a 5-point Likert scale ranging from Strongly Agree (4) to (0) Strongly Disagree.
Subjective Norms and Enabling Factors of Nail-Biting Among Children | one month
  The questionnaire includes ten yes/No questions divided into two categories. The subjective norms category consists of 8 items describing the external factors that influence children either to increase or quit their nails

CONTACTS AND LOCATIONS:
Overall Officials: Zohour I Rashwan, Professor, Principal Investigator — Alexandria University
Locations (1):
- Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zareipour MA, Mahmoodi H, Valizadeh R, Ghelichi Ghojogh M, Rezaie Moradali M, Zare F. Impact of an Educational Intervention Based on the BASNEF Model on Skin Cancer Preventive Behavior of College Students. Asian Pac J Cancer Prev. 2018 Oct 26;19(10):2717-2722. doi: 10.22034/APJCP.2018.19.10.2717. PMID 30360596
- [Background] Abd-Elsabour MAA, Hanafy RMH, Omar OM. Association between children's resilience and practising oral habits: a cross-sectional study. Br Dent J. 2023 Feb 17:1-5. doi: 10.1038/s41415-023-5565-7. Online ahead of print. PMID 36801961
- [Background] Gur K, Erol S, Incir N. The effectiveness of a nail-biting prevention program among primary school students. J Spec Pediatr Nurs. 2018 Jul;23(3):e12219. doi: 10.1111/jspn.12219. Epub 2018 May 24. PMID 29797491
- [Background] Ghanizadeh A, Shekoohi H. Prevalence of nail biting and its association with mental health in a community sample of children. BMC Res Notes. 2011 Apr 11;4:116. doi: 10.1186/1756-0500-4-116. PMID 21481256
- [Background] Ergun A, Toprak R, Sisman FN. Impact of a healthy nails program on nail-biting in Turkish schoolchildren: a controlled pretest-posttest study. J Sch Nurs. 2013 Dec;29(6):416-24. doi: 10.1177/1059840513481386. Epub 2013 Mar 14. PMID 23492878
- [Background] Silva LCD, Vedovello SAS, Vedovello Filho M, Meneghin MC, Ambrosano Bovi GM, Degan VV. Anxiety and oral habits as factors associated with malocclusion. Cranio. 2021 May;39(3):249-253. doi: 10.1080/08869634.2019.1633492. Epub 2019 Jun 23. PMID 31232226
- [Background] Baghchechi M, Pelletier JL, Jacob SE. Art of Prevention: The importance of tackling the nail biting habit. Int J Womens Dermatol. 2020 Sep 17;7(3):309-313. doi: 10.1016/j.ijwd.2020.09.008. eCollection 2021 Jun. PMID 32964094
- [Derived] Rashwan ZI, Darweesh HAM, Elsobky FA, Amer SAM, Nada MAA. BASNEF behavioral transformation: effect of empowerment program on children's knowledge, attitude, self-efficacy, and practice of nail biting. BMC Pediatr. 2025 Apr 22;25(1):312. doi: 10.1186/s12887-025-05450-w. PMID 40264049